CLINICAL TRIAL: NCT00368966
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in Spain
Brief Title: Study to Evaluate a 13-valent Pneumococcal Conjugate Vaccine in Infants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6096A1-501
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-07

CONDITIONS: Vaccines, Pneumococcal
Keywords: Pneumococcal; Pediatric; Vaccine
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- 2 (Active Comparator)
  Interventions: Biological: 7-valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine
  Arms: 1
Biological: 7-valent Pneumococcal Conjugate Vaccine
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate (13vPnC) vaccine compared to Prevenar (7vPnC), when given concomitantly with routine pediatric vaccinations in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month-old infants
* Available for the entire study period

Exclusion criteria:

* Previous vaccination with any vaccine before the start of the study
* Known contraindication to vaccination

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 619 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com
Locations (28):
- Spain (28):
  - A Coruña, A Coruna
  - Ferrol, A Coruna
  - Santiago de Compostela, A Coruna
  - Almería, Almeria
  - Argentona, Barcelona
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Sant Adrià de Besòs, Barcelona
  - Sant Cugat del Vallès, Barcelona
  - Bilbao, Bizkaia
  - A Coruña, La Coruna
  - Burela de Cabo, Lugo
  - Alcorcón, Madrid
  - Fuenlabrada, Madrid
  - Getafe, Madrid
  - Madrid, Madrid
  - Móstoles, Madrid
  - Parla, Madrid
  - Antequera, Malaga
  - Málaga, Malaga
  - Pamplona, Navarre
  - Ourense, Ourense
  - Vigo, Pontevedra
  - Seville, Sevilla
  - Burjassot, Valencia
  - L'Eliana, Valencia
  - Quart de Poblet, Valencia
  - Valencia, Valencia

REFERENCES:
- [Derived] Rodgers GL, Esposito S, Principi N, Gutierrez-Brito M, Diez-Domingo J, Pollard AJ, Snape MD, Martinon-Torres F, Gruber WC, Patterson S, Thompson A, Gurtman A, Paradiso P, Scott DA. Immune response to 13-valent pneumococcal conjugate vaccine with a reduced dosing schedule. Vaccine. 2013 Oct 1;31(42):4765-74. doi: 10.1016/j.vaccine.2013.08.009. Epub 2013 Aug 16. PMID 23965217
- [Derived] Gimenez-Sanchez F, Kieninger DM, Kueper K, Martinon-Torres F, Bernaola E, Diez-Domingo J, Steul K, Juergens C, Gurtman A, Giardina P, Liang JZ, Gruber WC, Emini EA, Scott DA; 501 and 006 study groups. Immunogenicity of a combination vaccine containing diphtheria toxoid, tetanus toxoid, three-component acellular pertussis, hepatitis B, inactivated polio virus, and Haemophilus influenzae type b when given concomitantly with 13-valent pneumococcal conjugate vaccine. Vaccine. 2011 Aug 11;29(35):6042-8. doi: 10.1016/j.vaccine.2011.06.026. Epub 2011 Jun 23. PMID 21704105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Spain from October 2006 to December 2006.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC: Participants received one single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with a combination vaccine diphtheria, tetanus, and pertussis (acellular) vaccine (DTPa), hepatitis B virus vaccine (HBV), inactivated poliovirus (IPV), and hemophilus influenza type b (Hib) vaccine (Infanrix hexa) and a meningococcal C conjugate vaccine (Meningitec) at 2 and 4 months. Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 6 months. Participants received one single 0.5 mL dose of 13vPnC coadministered with a combination vaccine measles, mumps, rubella live virus (MMR II) at 12 months. Participants received one single 0.5 mL dose of 13vPnC coadministered with DTPa, IPV, and Hib vaccine (Infanrix-IPV+Hib) and Meningitec at 15 months.
- 7vPnC: Participants received one single 0.5 milliliter (mL) dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with a combination vaccine diphtheria, tetanus, and pertussis (acellular) vaccine (DTPa), hepatitis B virus vaccine (HBV), inactivated poliovirus (IPV), and hemophilus influenza type b (Hib) vaccine (Infanrix hexa) and a meningococcal C conjugate vaccine (Meningitec) at 2 and 4 months. Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 6 months. Participants received one single 0.5 mL dose of 7vPnC coadministered with a combination vaccine measles, mumps, rubella live virus (MMR II) at 12 months. Participants received one single 0.5 mL dose of 7vPnC coadministered with DTPa, IPV, and Hib vaccine (Infanrix-IPV+Hib) and Meningitec at 15 months.
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 315 | 304
Vaccinated Dose 1 | 314 | 302 (1 randomized to 7vPnC but given 13vPnC vaccine; 1 was withdrawn before receiving 7vPnC vaccine)
Vaccinated Dose 2 | 307 (1 randomized but incorrectly given 7vPnC) | 298
Vaccinated Dose 3 | 301 | 296 (1 randomized but incorrectly given 13vPnC)
Completed | 299 | 294
Not Completed | 16 | 10
Not completed — Withdrawal by Subject | 11 | 6
Not completed — Protocol Violation | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Randomization error | 0 | 1
Not completed — Failed to meet eligibility criteria | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Failed to return | 1 | 0
Period: After Infant
Arm/Group | 13vPnC | 7vPnC
Started | 299 | 294
Completed | 293 | 289
Not Completed | 6 | 5
Not completed — Failed to return | 3 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 293 | 289
Completed | 292 | 286
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- 13vPnC: Subjects received 1 dose (0.5 mL) of 13vPnC together with 1 dose (0.5 mL) of each of the following concomitant vaccines: Infanrix hexa and Meningitec at 2 and 4 months. At 6 months subjects received 13vPnC and Infanrix hexa. At 12 months subjects received MMR II. At 15 months subjects received 13vPnC and Infanrix-IPV+Hib, Meningitec.
- 7vPnC: Subjects received 1 dose (0.5 mL) of 7vPnC together with 1 dose (0.5 mL) of each of the following concomitant vaccines: Infanrix hexa and Meningitec at 2 and 4 months. At 6 months subjects received 7vPnC and Infanrix hexa. At 12 months subjects received MMR II. At 15 months subjects received 7vPnC and Infanrix-IPV+Hib, Meningitec.
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 315 | 304 | 619
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.5) | 2.1 (0.5) | 2.1 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 152 | 300
  Male | 167 | 152 | 319

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Predefined Meningococcal C Serum Bactericidal Assay (SBA) Titer of ≥ 1:8, and a Predefined Antibody Level for Diphtheria in 13vPnC Group Relative to 7vPnC Group After 2-doses of the Infant Series
Description: Percentage of participants achieving predefined antibody threshold levels; greater than or equal to (≥) 1:8 for meningococcal C SBA titer and ≥ 0.10 or >=0.01 International Units Per Milliliter (IU/mL) for diphtheria along with the corresponding 95% Confidence Interval (CI) are presented.
Time Frame: One month after 2-doses of the infant series (5 months of age)
Population: Evaluable immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 2 and 4 months. Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 6 months (infant series). Participants received one single 0.5 mL dose of 13vPnC coadministered with MMR II at 12 months. Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months (toddler dose).
- 7vPnC: Participants received one single 0.5 mL dose of 7vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 2 and 4 months. Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 6 months (infant series). Participants received one single 0.5 mL dose of 7vPnC coadministered with MMR II at 12 months. Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months (toddler dose).
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 297 | 284
Percentage of Participants
  Meningococcal C ≥ 1:8 | 98.3 [96.1 to 99.5] | 98.9 [96.9 to 99.8]
  Diptheria ≥ 0.10 IU/mL | 95.9 [93.0 to 97.9] | 94.7 [91.4 to 97.0]
  Diptheria ≥ 0.01 IU/mL | 100.0 [98.8 to 100.0] | 100.0 [98.7 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Meningococcal C the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥ 1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) greater than (>) -10%; Difference = -0.6, 95% CI [-2.9 to 1.6]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Diphtheria the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥ 0.10 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lowest limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) > -10%; Difference = 1.2, 95% CI [-2.3 to 4.9]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Diphtheria the difference in percentage between the two groups (13vPnC - 7vPnC) at ≥ 0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.3 to 1.3]

2. Primary Outcome: Geometric Mean Titer (GMT) of Meningococcal C in 13vPnC Group Relative to 7vPnC Group After 2-doses of the Infant Series
Time Frame: One month after 2-doses of the infant series (5 months of age)
Population: The evaluable immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 2 and 4 months. Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 6 months (infant series). Participants received one single 0.5 mL dose of 13vPnC coadministered with MMR II at 12 months. Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months(toddler dose).
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 297 | 284
titer | 191.22 [167.72 to 218.02] | 266.19 [234.86 to 301.71]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Meningococcal C the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for immune response induced by Meningitec was declared if the lower bound of the 2-sided, 95% CI for the GMT ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.72, 95% CI [0.60 to 0.86]

3. Primary Outcome: Geometric Mean Antibody Concentration (GMC) for Diphtheria in 13vPnC Group Relative to 7vPnC Group After 2-doses of the Infant Series
Time Frame: One month after 2-doses of the infant series (5 months of age)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 296 | 284
IU/mL | 0.51 [0.47 to 0.57] | 0.63 [0.57 to 0.70]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Diphtheria the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for immune response induced by Meningitec was declared if the lower bound of the 2-sided, 95% CI for the GMC ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.81, 95% CI [0.70 to 0.94]

4. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were collected using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (Sig) (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (Mod) (2.5 to 7.0 cm); Severe (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5 mL dose of 13vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 2 months (infant series).
- 7vPnC Dose 1: Participants received one single 0.5 mL dose of 7vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 2 months (infant series).
- 13vPnC Dose 2: Participants received one single 0.5 mL dose of 13vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 4 months (infant series).
- 7vPnC Dose 2: Participants received one single 0.5 mL dose of 7vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 4 months (infant series).
- 13vPnC Dose 3: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 6 months (infant series).
- 7vPnC Dose 3: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 6 months (infant series).
- 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months (toddler dose).
- 7vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months (toddler dose).
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 314 | 300 | 306 | 298 | 301 | 295 | 293 | 289
percentage of participants
  Tenderness-Any (n=275,270,227,232,217,215,193,170) | 49.5 | 43.3 | 45.4 | 46.6 | 47.9 | 41.9 | 64.2 | 64.7
  Tenderness-Sig (n=247,250,192,203,181,171,136,118 | 2.8 | 2.8 | 4.2 | 3.9 | 6.1 | 0.0 | 5.9 | 6.8
  Swelling-Any (n=252,254,206,212,203,181,153,140) | 19.0 | 14.2 | 28.2 | 23.1 | 27.6 | 28.2 | 33.3 | 30.7
  Swelling-Mild (n=251,254,206,212,201,186,151,132) | 16.3 | 14.2 | 25.7 | 20.3 | 26.4 | 25.8 | 31.1 | 24.2
  Swelling-Mod (n=247,248,191,201,180,173,136,124) | 4.9 | 1.6 | 5.8 | 4.5 | 5.6 | 4.0 | 11.8 | 12.9
  Swelling-Severe(n=246,247,191,201,176,171,131,113) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Redness-Any (n=255,251,211,217,203,198,159,146) | 22.0 | 19.1 | 34.1 | 30.9 | 31.0 | 34.8 | 40.9 | 41.1
  Redness-Mild (n=254,251,210,215,203,195,157,141) | 20.1 | 18.3 | 32.4 | 30.2 | 29.1 | 33.3 | 35.0 | 37.6
  Redness-Mod (n=247,247,192,203,177,175,137,120) | 2.4 | 1.2 | 3.1 | 2.5 | 4.5 | 5.1 | 13.1 | 12.5
  Redness-Severe (n=246,247,191,201,176,171,131,113) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

5. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever [Fv] ≥ 37.5 degrees Celsius [C], fever ≥ 38 C but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased [Decr] appetite, irritability, increased [Incr] sleep, decreased sleep, hives, use of medication [Med] to treat symptoms [sx], and use of medication to prevent symptoms) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all subjects who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Dose 3 | 7vPnC Dose 3 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 314 | 300 | 306 | 298 | 301 | 295 | 293 | 289
percentage of participants
  Fv≥38°C, ≤39°C (n=262,253,213,223,198,196,162,145) | 30.5 | 24.5 | 40.4 | 41.7 | 34.3 | 38.3 | 38.9 | 44.8
  Fv>39°C, ≤40°C (n=249,247,194,204,177,174,135,118) | 0.8 | 0.8 | 2.6 | 2.5 | 5.6 | 5.2 | 8.1 | 6.8
  Fv >40°C (n=249,247,192,201,176,171,132,113) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.8 | 0.0
  Decr appetite (n=269,258,226,229,219,204,174,147) | 39.8 | 36.8 | 45.1 | 44.5 | 47.0 | 42.6 | 53.4 | 47.6
  Irritability (n=276,267,234,244,229,221,183,170) | 51.4 | 42.7 | 64.5 | 61.5 | 57.2 | 58.8 | 61.7 | 61.8
  Incr sleep (n=273,269,218,221,206,203,160,145) | 53.5 | 51.3 | 46.8 | 41.6 | 33.5 | 34.5 | 39.4 | 35.2
  Decr sleep (n=263,255,218,223,205,190,151,129) | 34.6 | 24.7 | 36.2 | 29.6 | 30.2 | 25.8 | 27.2 | 27.1
  Med-treat sx (n=267,256,232,243,216,209,176,163) | 50.6 | 46.9 | 60.3 | 61.3 | 55.6 | 55.5 | 59.7 | 60.1
  Med-prevent sx (n=269,258,231,237,222,211,178,159) | 49.1 | 47.7 | 58.4 | 58.6 | 56.3 | 53.6 | 59.6 | 61.6

6. Primary Outcome: Geometric Mean Antibody Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody in 13vPnC Group After the Second Dose and After the Third Dose of a 3-Dose Infant Series and After the Toddler Dose
Description: GMC as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes which are present in both 7vPnC and 13vPnC (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after infant series dose 2 (at 5 months of age) and dose 3 (at 7 months of age) and one month after the toddler dose (at 16 months of age)
Population: The evaluable immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- 13vPnC After Infant Series Dose 2: Participants received one single 0.5 mL dose of 13vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 2 and 4 months (infant series).
- 13vPnC After Infant Series Dose 3: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 6 months (infant series).
- 13vPnC After the Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months (toddler dose).
Arm/Group | 13vPnC After Infant Series Dose 2 | 13vPnC After Infant Series Dose 3 | 13vPnC After the Toddler Dose
Number analyzed (Participants) | 297 | 293 | 275
μg/mL
  Common Serotype - Serotype 4 (n=269,269,241) | 1.89 [1.70 to 2.10] | 2.33 [2.11 to 2.57] | 4.97 [4.42 to 5.58]
  Common Serotype - Serotype 6B (n=267,267,228) | 0.42 [0.37 to 0.47] | 3.88 [3.41 to 4.41] | 11.88 [10.57 to 13.35]
  Common Serotype - Serotype 9V (n=273,273,241) | 1.49 [1.34 to 1.66] | 1.71 [1.56 to 1.86] | 3.44 [3.12 to 3.80]
  Common Serotype - Serotype 14 (n=270,270,230) | 3.84 [3.37 to 4.37] | 6.17 [5.45 to 6.98] | 11.37 [10.17 to 12.71]
  Common Serotype - Serotype 18C (n=267,267,239) | 1.58 [1.40 to 1.78] | 2.29 [2.08 to 2.52] | 3.96 [3.55 to 4.43]
  Common Serotype - Serotype 19F (n=270,270,231) | 2.85 [2.53 to 3.21] | 2.64 [2.42 to 2.89] | 8.04 [7.07 to 9.14]
  Common Serotype - Serotype 23F (n=260,260,233) | 0.54 [0.47 to 0.62] | 2.15 [1.89 to 2.45] | 5.07 [4.50 to 5.71]
  Additional Serotype - Serotype 1 (n=268,268,235) | 1.90 [1.70 to 2.13] | 3.04 [2.73 to 3.38] | 4.79 [4.21 to 5.45]
  Additional Serotype - Serotype 3 (n=267,267,243) | 0.79 [0.72 to 0.87] | 0.97 [0.87 to 1.08] | 1.07 [0.95 to 1.20]
  Additional Serotype - Serotype 5 (n=261,261,234) | 0.99 [0.90 to 1.10] | 1.93 [1.74 to 2.13] | 3.90 [3.53 to 4.31]
  Additional Serotype - Serotype 6A (n=269,269,235) | 1.10 [0.97 to 1.25] | 3.16 [2.82 to 3.53] | 7.07 [6.35 to 7.87]
  Additional Serotype - Serotype 7F (n=268,268,242) | 1.85 [1.69 to 2.02] | 4.03 [3.70 to 4.40] | 5.78 [5.13 to 6.53]
  Additional Serotype - Serotype 19A (n=267,267,226) | 2.36 [2.10 to 2.66] | 3.07 [2.79 to 3.37] | 11.64 [10.43 to 13.00]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 4, the Geometric Mean fold Rise (GMFR) were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 1.23, 95% CI [1.13 to 1.35]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 6B the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Superiority or Other; Difference = 9.28, 95% CI [8.18 to 10.53]
Statistical Analysis 3: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 6B, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 1.15, 95% CI [1.05 to 1.25]
Statistical Analysis 4: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 14, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 1.61, 95% CI [1.41 to 1.83]
Statistical Analysis 5: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 18C, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 1.45, 95% CI [1.30 to 1.61]
Statistical Analysis 6: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 19F, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 0.93, 95% CI [0.83 to 1.03]
Statistical Analysis 7: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 23F, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 4.00, 95% CI [3.55 to 4.50]
Statistical Analysis 8: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 1, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 1.60, 95% CI [1.46 to 1.76]
Statistical Analysis 9: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 3, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 1.23, 95% CI [1.13 to 1.35]
Statistical Analysis 10: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 5, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 1.94, 95% CI [1.78 to 2.11]
Statistical Analysis 11: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 6A, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 2.87, 95% CI [2.58 to 3.20]
Statistical Analysis 12: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 7F, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 2.18, 95% CI [1.98 to 2.41]
Statistical Analysis 13: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 19A, the GMFR were calculated using all participants with available data from both 13vPnC After Infant Series Dose 2 and 13vPnC After Infant Series Dose 3 blood draws; Test type: Superiority or Other; Difference = 1.30, 95% CI [1.18 to 1.44]

7. Primary Outcome: Percentage of Participants Achieving Predefined Antibody Levels for Pertussis, Diphtheria, Tetanus, and Poliovirus in 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series and the Toddler Dose
Description: Percentage of participants achieving predefined antibody threshold levels with the corresponding 95% CI for each concomitant antigen (pertussis antigens including Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA), and Pertactin (PRN); diphtheria; tetanus; and poliovirus types 1, 2, and 3) are presented.
Time Frame: One month after the 3-dose infant series (7 months of age) and the toddler dose (16 months of age)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC After Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 6 months (infant series).
- 7vPnC After Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 6 months (infant series).
- 7vPnC After the Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months.
Arm/Group | 13vPnC After Infant Series | 7vPnC After Infant Series | 13vPnC After the Toddler Dose | 7vPnC After the Toddler Dose
Number analyzed (Participants) | 293 | 286 | 275 | 270
percentage of participants
  Pertussis, PT ≥ 5.0 EU/mL | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 99.6 [98.0 to 100.0] | 99.6 [97.9 to 100.0]
  Pertussis, PT (Infant ≥ 20; Toddler ≥ 11) EU/mL | 93.2 [89.7 to 95.8] | 95.1 [91.9 to 97.3] | 94.9 [91.6 to 97.2] | 96.3 [93.3 to 98.2]
  Pertussis, FHA ≥ 5.0 EU/mL | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.6 to 100.0]
  Pertussis, FHA ≥ 7.82 EU/mL | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.6 to 100.0]
  Pertussis, FHA (Infant ≥ 64; Toddler ≥ 99) EU/mL | 93.9 [90.5 to 96.3] | 95.1 [91.9 to 97.3] | 94.5 [91.1 to 96.9] | 95.1 [91.8 to 97.4]
  Pertussis, PRN ≥ 5 EU/mL | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.6 to 100.0]
  Pertussis, PRN (Infant ≥ 39; Toddler ≥ 69) EU/mL | 94.5 [91.3 to 96.8] | 95.1 [91.9 to 97.3] | 93.5 [89.9 to 96.1] | 95.2 [91.9 to 97.4]
  Diptheria ≥ 0.10 IU/mL | 99.3 [97.5 to 99.9] | 100.0 [98.7 to 100.0] | 99.2 [97.2 to 99.9] | 100.0 [98.5 to 100.0]
  Diptheria ≥ 0.01 IU/mL | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.5 to 100.0]
  Tetanus ≥ 0.10 IU/mL | 98.6 [96.3 to 99.6] | 98.2 [95.8 to 99.4] | 98.6 [95.9 to 99.7] | 97.8 [94.9 to 99.3]
  Tetanus ≥ 0.01 IU/mL | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.3 to 100.0] | 100.0 [98.4 to 100.0]
  Poliovirus, Type 1 ≥ 1:8 | 100.0 [98.7 to 100.0] | 100.0 [98.7 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0]
  Poliovirus, Type 2 ≥ 1:8 | 100.0 [98.7 to 100.0] | 99.3 [97.5 to 99.9] | 100.0 [98.6 to 100.0] | 99.6 [97.8 to 100.0]
  Poliovirus, Type 3 ≥ 1:8 | 100.0 [98.7 to 100.0] | 99.6 [98.0 to 100.0] | 100.0 [98.6 to 100.0] | 100.0 [98.6 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Pertussis, PT the difference in percentage between the two groups (13vPnC - 7vPnC) at 5.0 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.3 to 1.3]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Pertussis, PT the difference in percentage between the two groups (13vPnC - 7vPnC) at 20 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = -1.9, 95% CI [-6.0 to 2.0]
Statistical Analysis 3: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Pertussis, FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 5.0 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.3 to 1.3]
Statistical Analysis 4: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Pertussis, FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 7.82 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.3 to 1.3]
Statistical Analysis 5: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Pertussis, FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 64 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = -1.3, 95% CI [-5.2 to 2.6]
Statistical Analysis 6: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Pertussis, PRN the difference in percentage between the two groups (13vPnC - 7vPnC) at 5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.3 to 1.3]
Statistical Analysis 7: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Pertussis, PRN the difference in percentage between the two groups (13vPnC - 7vPnC) at 39 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = -0.6, 95% CI [-4.4 to 3.2]
Statistical Analysis 8: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.7 to 1.7]
Statistical Analysis 9: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis, PT the difference in percentage between the two groups (13vPnC - 7vPnC) at 11 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = -1.4, 95% CI [-5.1 to 2.2]
Statistical Analysis 10: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 7, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 11: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 7, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 12: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis, FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 99 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = -0.6, 95% CI [-4.6 to 3.3]
Statistical Analysis 13: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 7, analysis 6]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI [-1.4 to 1.4]
Statistical Analysis 14: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Pertussis, PRN the difference in percentage between the two groups (13vPnC - 7vPnC) at 69 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = -1.7, 95% CI [-5.8 to 2.3]
Statistical Analysis 15: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Diphtheria the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.10 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = -0.7, 95% CI 2-sided [-2.5 to 0.7]
Statistical Analysis 16: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Diphtheria the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI 2-sided [-1.3 to 1.3]
Statistical Analysis 17: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 7, analysis 15]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = -0.8, 95% CI 2-sided [-2.8 to 0.8]
Statistical Analysis 18: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; [analysis description as in outcome 7, analysis 16]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI 2-sided [-1.5 to 1.5]
Statistical Analysis 19: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Tetanus the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.10 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.4, 95% CI 2-sided [-2.1 to 2.9]
Statistical Analysis 20: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Tetanus the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI 2-sided [-1.3 to 1.3]
Statistical Analysis 21: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Tetanus the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.10 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.8, 95% CI 2-sided [-2.1 to 3.8]
Statistical Analysis 22: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Tetanus the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.01 IU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI 2-sided [-1.8 to 1.7]
Statistical Analysis 23: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Poliovirus Type 1 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI 2-sided [-1.4 to 1.3]
Statistical Analysis 24: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Poliovirus Type 2 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.7, 95% CI 2-sided [-0.6 to 2.6]
Statistical Analysis 25: Comparison: 13vPnC After Infant Series vs 7vPnC After Infant Series; For Poliovirus Type 3 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.4, 95% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 26: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Poliovirus Type 1 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI 2-sided [-1.5 to 1.5]
Statistical Analysis 27: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Poliovirus Type 2 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.4, 95% CI 2-sided [-1.1 to 2.2]
Statistical Analysis 28: Comparison: 13vPnC After the Toddler Dose vs 7vPnC After the Toddler Dose; For Poliovirus Type 3 the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Difference = 0.0, 95% CI 2-sided [-1.5 to 1.5]

8. Primary Outcome: Geometric Mean Titers (GMT) for Poliovirus in 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series and the Toddler Dose
Time Frame: One month after the 3-dose infant series (7 months of age) and the toddler dose (16 months of age)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 7vPnC After Infant Series Dose 3: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 6 months (infant series).
- 7vPnC Afte the Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months (toddler dose).
Arm/Group | 13vPnC After Infant Series Dose 3 | 7vPnC After Infant Series Dose 3 | 13vPnC After the Toddler Dose | 7vPnC Afte the Toddler Dose
Number analyzed (Participants) | 293 | 286 | 275 | 270
titer
  Poliovirus Type 1 | 436.98 [378.21 to 504.88] | 436.15 [378.17 to 503.02] | 1057.40 [939.06 to 1190.70] | 1286.70 [1131.00 to 1463.80]
  Poliovirus Type 2 | 266.34 [227.84 to 311.36] | 281.85 [240.04 to 330.94] | 1032.30 [912.96 to 1167.10] | 1141.10 [992.96 to 1311.40]
  Poliovirus Type 3 | 897.67 [766.30 to 1051.60] | 943.95 [806.71 to 1104.50] | 2571.10 [2249.40 to 2938.90] | 2410.80 [2106.70 to 2758.80]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For Poliovirus Type 1 the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the GMT ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 1.00, 95% CI [0.82 to 1.23]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For Poliovirus Type 2 the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; Ratio = 0.94, 95% CI [0.76 to 1.18]
Statistical Analysis 3: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For Poliovirus Type 3 the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; Ratio = 0.95, 95% CI [0.76 to 1.19]
Statistical Analysis 4: Comparison: 13vPnC After the Toddler Dose; For Poliovirus Type 1 the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; Ratio = 0.82, 95% CI [0.69 to 0.98]
Statistical Analysis 5: Comparison: 13vPnC After the Toddler Dose vs 7vPnC Afte the Toddler Dose; For Poliovirus Type 2 the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; Ratio = 0.90, 95% CI [0.75 to 1.09]
Statistical Analysis 6: Comparison: 13vPnC After the Toddler Dose vs 7vPnC Afte the Toddler Dose; For Poliovirus Type 3 the GMT ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; Ratio = 1.07, 95% CI [0.88 to 1.29]

9. Primary Outcome: Geometric Mean Antibody Concentrations (GMC) for Diphtheria and Tetanus in 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series and the Toddler Dose
Time Frame: One month after the 3-dose infant series (7 months of age) and the toddler dose (16 months of age)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 13vPnC After Infant Series Dose 3 | 7vPnC After Infant Series Dose 3 | 13vPnC After the Toddler Dose | 7vPnC Afte the Toddler Dose
Number analyzed (Participants) | 293 | 286 | 275 | 270
IU/mL
  Diphtheria | 1.19 [1.08 to 1.30] | 1.40 [1.28 to 1.53] | 3.00 [2.65 to 3.40] | 3.51 [3.08 to 3.99]
  Tetanus | 0.90 [0.80 to 1.01] | 0.87 [0.79 to 0.97] | 1.63 [1.38 to 1.91] | 1.45 [1.24 to 1.69]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For diphtheria toxoid the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the GMC ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.85, 95% CI [0.75 to 0.96]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For Tetanus the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 1.03, 95% CI [0.88 to 1.20]
Statistical Analysis 3: Comparison: 13vPnC After the Toddler Dose vs 7vPnC Afte the Toddler Dose; For diphtheria toxoid the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 0.86, 95% CI [0.71 to 1.02]
Statistical Analysis 4: Comparison: 13vPnC After the Toddler Dose vs 7vPnC Afte the Toddler Dose; For Tetanus the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 1.12, 95% CI [0.90 to 1.40]

10. Primary Outcome: Geometric Mean Antibody Concentrations (GMC) for Pertussis in 13vPnC Group Relative to 7vPnC Group After the 3-dose Infant Series and the Toddler Dose
Description: GMCs with the corresponding 95% CI for each concomitant antigen pertussis antigens (PT, FHA, PRN, and FIM) as measured by EU/mL are presented.
Time Frame: One month after the 3-dose infant series (7 months of age) and the toddler dose (16 months of age)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 13vPnC After Infant Series Dose 3 | 7vPnC After Infant Series Dose 3 | 13vPnC After the Toddler Dose | 7vPnC Afte the Toddler Dose
Number analyzed (Participants) | 293 | 286 | 275 | 270
EU/mL
  Pertussis PT | 51.51 [47.94 to 55.34] | 50.13 [46.80 to 53.70] | 36.13 [32.84 to 39.74] | 36.01 [32.94 to 39.37]
  Pertussis FHA | 179.04 [165.34 to 193.87] | 166.77 [155.20 to 179.20] | 347.96 [316.46 to 382.59] | 345.89 [315.14 to 379.65]
  Pertussis PRN | 141.39 [129.66 to 154.17] | 135.06 [123.56 to 147.63] | 232.96 [211.42 to 256.69] | 261.58 [237.29 to 288.36]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For Pertussis PT the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 1.03, 95% CI [0.93 to 1.13]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For Pertussis FHA the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 1.07, 95% CI [0.96 to 1.20]
Statistical Analysis 3: Comparison: 13vPnC After Infant Series Dose 3 vs 7vPnC After Infant Series Dose 3; For Pertussis PRN the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 1.05, 95% CI [0.92 to 1.18]
Statistical Analysis 4: Comparison: 13vPnC After the Toddler Dose vs 7vPnC Afte the Toddler Dose; For Pertussis PT the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 1.00, 95% CI [0.88 to 1.14]
Statistical Analysis 5: Comparison: 13vPnC After the Toddler Dose vs 7vPnC Afte the Toddler Dose; For Pertussis FHA the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 1.01, 95% CI [0.88 to 1.15]
Statistical Analysis 6: Comparison: 13vPnC After the Toddler Dose vs 7vPnC Afte the Toddler Dose; For Pertussis PRN the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; Ratio = 0.89, 95% CI [0.78 to 1.02]

11. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥ 0.35 Microgram Per Milliliter (μg/mL) in 13vPnC Group After the Second Dose and After the Third Dose of a 3-Dose Infant Series and After the Toddler Dose
Description: Percentages of participants achieving World Health Organization (WHO) predefined antibody threshold ≥ 0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes, present in both 13vPnC and 7vPnC (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- 13vPnC After Infant Series Dose 2: Participants received one single 0.5 mL dose of 13vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 4 months (infant series).
Arm/Group | 13vPnC After Infant Series Dose 2 | 13vPnC After Infant Series Dose 3 | 13vPnC After the Toddler Dose
Number analyzed (Participants) | 297 | 293 | 275
Percentage of Participants
  Common Serotype - Serotype 4 | 96.7 [93.7 to 98.5] | 98.9 [96.8 to 99.8] | 99.2 [97.0 to 99.9]
  Common Serotype - Serotype 6B | 57.3 [51.1 to 63.3] | 98.5 [96.2 to 99.6] | 99.6 [97.6 to 100.0]
  Common Serotype - Serotype 9V | 91.9 [88.1 to 94.9] | 99.3 [97.4 to 99.9] | 100.0 [98.5 to 100.0]
  Common Serotype - Serotype 14 | 98.5 [96.3 to 99.6] | 97.4 [94.7 to 99.0] | 100.0 [98.4 to 100.0]
  Common Serotype - Serotype 18C | 91.8 [87.8 to 94.8] | 98.1 [95.7 to 99.4] | 99.6 [97.7 to 100.0]
  Common Serotype - Serotype 19F | 97.8 [95.2 to 99.2] | 99.3 [97.3 to 99.9] | 99.6 [97.6 to 100.0]
  Common Serotype - Serotype 23F | 68.1 [62.0 to 73.7] | 94.6 [91.1 to 97.0] | 99.1 [96.9 to 99.9]
  Additional Serotype - Serotype 1 | 96.3 [93.2 to 98.2] | 99.3 [97.3 to 99.9] | 98.7 [96.3 to 99.7]
  Additional Serotype - Serotype 3 | 88.0 [83.5 to 91.7] | 90.3 [86.1 to 93.5] | 92.2 [88.1 to 95.2]
  Additional Serotype - Serotype 5 | 87.4 [82.7 to 91.1] | 97.3 [94.6 to 98.9] | 99.1 [96.9 to 99.9]
  Additional Serotype - Serotype 6A | 84.4 [79.5 to 88.5] | 97.4 [94.7 to 98.9] | 99.1 [97.0 to 99.9]
  Additional Serotype - Serotype 7F | 98.5 [96.2 to 99.6] | 100.0 [98.6 to 100.0] | 98.8 [96.4 to 99.7]
  Additional Serotype - Serotype 19A | 98.1 [95.7 to 99.4] | 99.6 [97.9 to 100.0] | 100.0 [98.4 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 4, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 2.2, 95% CI [0.1 to 4.4]
Statistical Analysis 2: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 6B, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 41.2, 95% CI [34.9 to 46.9]
Statistical Analysis 3: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 9V, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 7.3, 95% CI [4.1 to 10.4]
Statistical Analysis 4: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 14, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = -1.1, 95% CI [-3.4 to 1.2]
Statistical Analysis 5: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 18C, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 6.4, 95% CI [3.1 to 9.5]
Statistical Analysis 6: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 19F, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 1.5, 95% CI [-0.4 to 3.4]
Statistical Analysis 7: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 23F, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 26.5, 95% CI [20.7 to 31.9]
Statistical Analysis 8: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 1, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 3.0, 95% CI [0.8 to 5.1]
Statistical Analysis 9: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 3, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 2.2, 95% CI [-1.8 to 6.3]
Statistical Analysis 10: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 5, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 10.0, 95% CI [5.9 to 13.9]
Statistical Analysis 11: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 6A, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 13.0, 95% CI [8.6 to 17.2]
Statistical Analysis 12: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 7F, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 1.5, 95% CI [-0.1 to 3.1]
Statistical Analysis 13: Comparison: 13vPnC After Infant Series Dose 2 vs 13vPnC After Infant Series Dose 3; For serotype 19A, the difference in percentages between the two groups (13vPnC After Infant Series Dose 2 - 13vPnC After Infant Series Dose 3) was calculated; Test type: Superiority or Other; Difference = 1.5, 95% CI [-0.4 to 3.4]

ADVERSE EVENTS:
Groups:
- 13vPnC Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 2 and 4 months, assessment was done approximately one month after dose 2 at 5 months of age.
- 7vPnC Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with a combination vaccine Infanrix hexa and Meningitec at 2 and 4 months, assessment was done approximately one month after dose 2 at 5 months of age.
- 13vPnC Post-Infant Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix hexa at 6 months (infant series), assessment was done approximately one month after dose 3 at 7 months of age.
- 7vPnC Post-Infant Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix hexa at 6 months, assessment was done approximately one month after dose 3 at 7 months of age.
- 13vPnC Toddler Series: Participants received one single 0.5 mL dose of 13vPnC coadministered with MMR II at 12 months. Participants received one single 0.5 mL dose of 13vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months (toddler dose). Assessment was done approximately one month after toddler dose at 16 months of age.
- 7vPnC Toddler Series: Participants received one single 0.5 mL dose of 7vPnC coadministered with MMR II at 12 months. Participants received one single 0.5 mL dose of 7vPnC coadministered with Infanrix-IPV+Hib and Meningitec at 15 months (toddler dose). Assessment was done approximately one month after toddler dose at 16 months of age.
- 13vPnC 6-Month Follow-up: Assessment was done approximately 6 months after 13vPnC toddler dose at 21 months of age.
- 7vPnC 6-Month Follow-up: Assessment was done approximately 6 months after 7vPnC toddler dose at 21 months of age.
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC Post-Infant Series | 7vPnC Post-Infant Series | 13vPnC Toddler Series | 7vPnC Toddler Series | 13vPnC 6-Month Follow-up | 7vPnC 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 16/314 | 16/300 | 16/314 | 16/300 | 3/291 | 1/284 | 3/312 | 6/299
Other Adverse Events (participants affected / at risk) | 151/314 | 156/300 | 7/314 | 10/300 | 124/291 | 110/284 | 3/312 | 2/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=314) | 7vPnC Infant Series (N=300) | 13vPnC Post-Infant Series (N=314) | 7vPnC Post-Infant Series (N=300) | 13vPnC Toddler Series (N=291) | 7vPnC Toddler Series (N=284) | 13vPnC 6-Month Follow-up (N=312) | 7vPnC 6-Month Follow-up (N=299)
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Congenital nystagmus (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fontanelle bulging (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 0
Gastroenteritis rotavirus (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Gastroenteritis salmonella (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scaphocephaly (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden infant death syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 12/247 | 4/248 | 16/136 | 16/124 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=314) | 7vPnC Infant Series (N=300) | 13vPnC Post-Infant Series (N=314) | 7vPnC Post-Infant Series (N=300) | 13vPnC Toddler Series (N=291) | 7vPnC Toddler Series (N=284) | 13vPnC 6-Month Follow-up (N=312) | 7vPnC 6-Month Follow-up (N=299)
Hip dysplasia (Congenital, familial and genetic disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Double ureter (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypospadias (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Strabismus congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 10 | 10 | 0 | 1 | 9 | 3 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Conjuctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 5 | 1 | 0 | 5 | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 4 | 0 | 0 | 5 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 20 | 16 | 0 | 0 | 8 | 4 | 0 | 0
Irritability (General disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Milk allergy (Immune system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 53 | 47 | 0 | 0 | 15 | 12 | 0 | 0
Bronchiolitis (Infections and infestations) | 32 | 35 | 0 | 0 | 1 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 25 | 23 | 0 | 2 | 11 | 16 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 8 | 6 | 0 | 1 | 1 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 23 | 33 | 0 | 1 | 10 | 9 | 0 | 0
Gastroenteritis (Infections and infestations) | 19 | 22 | 0 | 0 | 16 | 15 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 5 | 7 | 0 | 0 | 6 | 6 | 0 | 0
Respiratory tract infection (Infections and infestations) | 9 | 2 | 0 | 0 | 5 | 4 | 0 | 0
Otitis media (Infections and infestations) | 3 | 6 | 0 | 0 | 4 | 5 | 0 | 0
Tonsillitis (Infections and infestations) | 3 | 3 | 0 | 0 | 2 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 4 | 1 | 0 | 0 | 1 | 3 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 3 | 0 | 0 | 2 | 3 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dacryocystitis (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral skin infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 | 9 | 0 | 0 | 1 | 0 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0 | 0 | 3 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Penis disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular retraction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exposure to communicable disease (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 136/275 | 117/270 | 0/0 | 0/0 | 124/193 | 110/170 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 103/227 | 108/232 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 104/217 | 90/215 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 7/247 | 7/250 | 0/0 | 0/0 | 8/136 | 8/118 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 8/192 | 8/203 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 11/181 | 0/171 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)
Induration (Any) (Skin and subcutaneous tissue disorders) | 48/252 | 36/254 | 0/0 | 0/0 | 51/153 | 43/140 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (any)=present at site of vaccination.
Induration (Any) (Skin and subcutaneous tissue disorders) | 58/206 | 49/212 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)
Induration (Any) (Skin and subcutaneous tissue disorders) | 56/203 | 53/188 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 41/251 | 36/254 | 0/0 | 0/0 | 47/151 | 32/132 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (Mild) (Skin and subcutaneous tissue disorders) | 53/206 | 43/212 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 53/201 | 48/186 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 12/247 | 4/248 | 0/0 | 0/0 | 16/136 | 16/124 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 11/191 | 9/201 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 10/180 | 7/173 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/246 | 0/247 | 0/0 | 0/0 | 0/131 | 0/113 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/191 | 0/201 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/176 | 0/171 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 56/255 | 48/251 | 0/0 | 0/0 | 65/159 | 60/146 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (any)=present at site of vaccination.
Erythema (Any) (Skin and subcutaneous tissue disorders) | 72/211 | 67/217 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 63/203 | 69/198 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (any)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 51/254 | 46/251 | 0/0 | 0/0 | 55/157 | 53/141 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 68/210 | 65/215 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 59/203 | 65/195 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (mild)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 6/247 | 3/247 | 0/0 | 0/0 | 18/137 | 15/120 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 6/192 | 5/203 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 8/177 | 9/175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (moderate)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/246 | 0/247 | 0/0 | 0/0 | 0/131 | 0/113 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/191 | 0/201 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/176 | 0/171 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (severe)
Fever ≥38°C but ≤39°C (General disorders) | 80/262 | 62/253 | 0/0 | 0/0 | 63/162 | 65/145 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but ≤39°C (General disorders) | 86/213 | 93/223 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but ≤39°C (General disorders) | 68/198 | 75/196 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38 degrees C but ≤39 degrees C
Fever >39°C but ≤40°C (General disorders) | 2/249 | 2/247 | 0/0 | 0/0 | 11/135 | 8/118 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but ≤40°C (General disorders) | 5/194 | 5/204 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but ≤40°C (General disorders) | 10/177 | 9/174 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39 degrees C but ≤40 degrees C
Fever >40°C (General disorders) | 0/249 | 0/247 | 0/0 | 0/0 | 1/132 | 0/113 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40 degrees C
Fever >40°C (General disorders) | 0/192 | 0/201 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40 degrees C
Fever >40°C (General disorders) | 0/176 | 0/171 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40 degrees C
Decreased appetite (General disorders) | 107/269 | 95/258 | 0/0 | 0/0 | 93/174 | 70/147 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 102/226 | 102/229 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 103/219 | 87/204 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 142/276 | 114/267 | 0/0 | 0/0 | 113/183 | 105/170 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 151/234 | 150/244 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 131/229 | 130/221 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 146/273 | 138/269 | 0/0 | 0/0 | 63/160 | 51/145 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 102/218 | 92/221 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 69/206 | 70/203 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 91/263 | 63/255 | 0/0 | 0/0 | 41/151 | 35/129 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 79/218 | 66/223 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 62/205 | 49/190 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 3 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.